CLINICAL TRIAL: NCT05862571
Title: Screening Instruments for Measuring Visual Symptoms in Victims of Concussion
Acronym: VISCOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: IT University of Copenhagen (Other); The Danish Victims Fund (Other Government); Synoptik-Fonden (Unknown); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Hana Malá Rytter, Head of the Danish Concussion Center, Associate Professor at University of Copenhagen and Neuropsychologist at Bispebjerg Hospital, Bispebjerg Hospital
Other Study IDs: VISCOM
Record Dates: First submitted 2023-03-23; First posted 2023-05-17 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Brain Concussion; mTBI - Mild Traumatic Brain Injury
Keywords: mTBI; Ocular Motility Disorders; Oculomotor Disorder; Mild Traumatic Brain Injury; Concussion; Mild Concussion; Eye tracking; Questionnaire
MeSH Terms: conditions — Brain Concussion; Ocular Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild traumatic brain injury group: Consist of patients who have been diagnosed with mTBI by a doctor at an emergency room or in general practice. The patients must still have symptoms related to their trauma ≥ 2 months and ≤ 24 months after trauma origin. They must not have received any vision therapy from an optometrist in relation to resent mTBI.
- Non-injured group: The control group will primarily consist of relatives of the individuals with mTBI, preferably a partner or a sibling. The subjects in the control group have to meet the same inclusion and exclusion criteria as the mTBI group, except that they must not be diagnosed with mild traumatic brain injury.

SUMMARY:
Visual dysfunction after mild traumatic brain injury (mTBI) is common but often remain undiscovered during longer periods of time. No valid, reliable and easy-to-use screening instrument for uncovering visual dysfunction exists. Furthermore, it is unknown whether optometric measurements currently used in assessing vision problems are consistent with patients' subjective complaints experienced in everyday life. A better understanding of patients' visual challenges combined with objective measurements, will contribute to a better and more efficient diagnostic investigation and treatment.

The aim of this study is to get a better understanding of patients who are suffering from visual dysfunction after mTBI. This understanding will be gained by:

1. developing and validating a questionnaire for uncovering subjective visual complaints in subjects with mTBI.
2. developing eye tracking based screening tools applicable both in- and outside of optometry clinics
3. examining relationships between self-reported data, eye tracking measurements and optometric measurements.

The study will consist of N = 200 subjects. N = 100 of the subjects are suffering from mTBI (commotio group). The second group N = 100 is the non-injured group that preferably will consist of relatives to the subjects in the commotio group. The subjects in both groups have to answer the questionnaires regarding subjective visual complains, undergo optometric tests and undergo eye tracking measurements.

ELIGIBILITY:
Inclusion Criteria:

Individuals may be included if they:

* are adults between the ages 18 and 67
* have been diagnosed with mTBI by a doctor (emergency room or general practice) either exclusively or with another diagnosis e.g. fracture, neck trauma (doesn't apply to control group)
* can read and understand Danish
* continuously have symptoms related to trauma ≥ 2 months and ≤ 24 months after trauma origin (doesn't apply to control group)
* have best corrected visus at 0.8 or better in both eyes at distance and at near
* have given informed consent and willingness to participate in the study

Exclusion Criteria:

The following will be excluded if individuals:

* are diagnosed with one of the following neurological disorders: severe head trauma, brain tumor, Parkinson's disease, multiple sclerosis, dementia
* are diagnosed with a current active psychiatric disorder
* are diagnosed with one of the following somatic disorders which are unregulated: diabetes mellitus, metabolic disorders
* have a verified alcohol or drug abuse
* have amblyopia (that is, two lines difference or more in best corrected visus between the two eyes)
* have other visual problems such as constant strabismus, a history of strabismus surgery, congenital nystagmus and recognized eye illnesses such as glaucoma, age- related macular degeneration (AMD)
* have received vision therapy by an optometrist in relation to resent mTBI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects (N=200) will be recruited through 5 optometric clinics on Zealand, DK. The objective is to recruit 100 individuals with mTBI and 100 individuals without mTBI (control group). The control group will consist of relatives of the individuals with mTBI, preferably a partner or a sibling.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
VISCOM Questionnaire | Estimated duration: 20 minutes
  Development and validation of the VISCOM questionnaire consisting of 42 times and establishing a cut-off score, with the aim of uncovering subjective visual symptoms after mTBI. The patients can score their visual symptoms on a Likert scale from 1-5, where one is "never" and five is "always". The higher score the more severe symptoms. The patient symptom score will be compared to the control group symptom score.

SECONDARY OUTCOMES:
The Rivermead Post Concussion Symptoms Questionnaire (RPQ) | Estimated duration in total: 5 minutes
  Valid questionnaire consisting 16 items, assessing symptoms after mTBI. The patients can score their visual symptoms from 1-5, one is "not experienced at all" and five is "a severe problem". The higher score, the more server symptoms.
Vergence facility | Estimated duration in total: 2 minutes
  A test of the eyes ability to converge and diverge using a 12 pd base out and 3 pd base in vergence flipper. The result is measured in cycles per minute, using a vertical line of letters 0,4/0,6 ≤ 35 years, and 0,4/1,0 >35 years.
Fusional vergence at near | Estimated duration in total: 2 minutes
  A test of the eyes ability to maintain fusion at 0,4 meter using rotary prism, both positive and negative fusional vergence. The result is measured in prism diopters using a vertical line of letters 0,4/0,6.
Monocular amplitude of accommodation | Estimated duration in total: 2 minutes
  A test of the eyes ability to accommodate using the Accommodation and Near Point Rule. The result is measured in cm using a vertical line with letters 0,4/0,6 with patients ≤ 35 years. The test is done separately with right and left eye.
Monocular accommodation facility | Estimated duration in total: 2 minutes
  A test of the eyes ability to accommodate and relax using a using a ± 2.00 accommodative flipper. The result is measured in cycles per minute, using a vertical line of letters 0,4/0,6 patients ≤ 35 years.
Horizontal and vertical phoria | Estimated duration in total: 2 minutes
  A test of the eyes natural alignment or misalignment using Modified Thorington Test measured in prism diopters at 6 meter and 0,4 meter.
Near point of convergence | Estimated duration in total: 5 minutes
  A test of the eyes ability to converge using the Accommodation and Near Point Rule. The result is measured in cm using a vertical line with letters 0,4/0,6 ≤ 35 years, and 0,4/1,0 >35 years. The test is repeated twice in the optometry clinic and twice using an eye-tracking setup.
Saccadic eye movement | Estimated duration in total: 10 minutes
  A test of the of saccades using 3 test cards and one demonstration card, in the optometry clinic and also using an eye-tracking setup. The result is measured in seconds and errors in total.
Reaction test | Estimated duration in total: 5 minutes
  An eye-tracking test of the participant's reaction time for a visual target appearing after a random delay. The result is measured as delay from the target appears to the following reactions: eye movement initiation, target fixation. Additionally, the accuracy of the initial fixation is measured. The test is repeated 24 times with delays drawn from three normal distributions. The delays are identical between participants.
Pattern test | Estimated duration in total: 5 minutes
  An eye-tracking test of the participant's ability to follow a moving circular target placed in a grid of identical moving targets. The target's position and direction of movement is indicated before the test is started. The result is measured as average fixation accuracy over the test period. The test is repeated 24 times with varying movement speed, direction, and target size.
Saccade test | Estimated duration in total: 5 minutes
  An eye-tracking of the participant's ability to quickly move their eyes between two targets in a given timeframe. The targets are circular and vary in size and position for each test repetition. The result is measured in number of correct saccades between the targets as well as the average fixation error (fixation distance outside target).
Smooth pursuit test | Estimated duration in total: 5 minutes
  An eye-tracking of the participant's ability to follow a small circular target's movements across a screen at various speeds and movement patterns. The test is repeated a total of 25 times comprised of 5 movement speeds for each of 5 patterns (horizontal line, vertical line, two diagonal lines, circle). The result is measured as average target deviation, number and duration of blinks, and number and amplitude of saccadic movements.

OTHER OUTCOMES:
Nystagmus test | Estimated duration in total: 5 minutes
  An eye-tracking test of the participant's ability to hold each eye still in an outward position for a duration of 10 seconds. The result is measured in the number and amplitude of saccadic movements over the time period.
Stereopsis | Estimated duration in total: 2 minutes.
  A test and evaluation of the eyes depth perception using polaroid glasses and Random Dot Stereotest. The result is measured in seconds of arc.
Vectogram no.12 | Estimated duration in total: 2 minutes
  The Vectogram no. 12 test is done at 0,4 meter, while the patient is reporting how exhausting the test is on a score from 1-5, where one is "easy and without trouble" and 5 is "unbearable exhausting". The result from the Vectogram no. 12 is measured in prism diopters.

CONTACTS AND LOCATIONS:
Overall Officials: Hana M Rytter, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No